CLINICAL TRIAL: NCT02503254
Title: A Randomized, Controlled, Open-label, 2-arm Parallel Group, Single Center Study to Demonstrate Reductions in Exposure to Selected Smoke Constituents in Healthy Smokers Switching to the Carbon Heated Tobacco Product 1.0 (CHTP 1.0) Compared to Continuing to Use Conventional Cigarettes During 5 Days in Confinement.
Brief Title: Reduced Exposure Study Using CHTP 1.0 During 5 Days in Confinement.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P2R-REXC-06-EU; P2R-REXC-06-EU (Other: Philip Morris Products S.A.)
Record Dates: First submitted 2015-07-17; First posted 2015-07-20 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Smoking
Keywords: Smoking; Modified risk tobacco product; Conventional cigarette; Reduced exposure; Confinement; Carbon Heated Tobacco Product
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHTP 1.0 (Experimental): Ad libitum use of the Carbon Heated Tobacco Product 1.0 (CHTP 1.0) for 5 days in confinement
  Interventions: Other: CHTP 1.0
- Conventional cigarette (CC) (Active Comparator): Ad libitum use of subject's own preferred brand of CC for 5 days in confinement
  Interventions: Other: Conventional Cigarette (CC)

INTERVENTIONS:
Other: CHTP 1.0 — CHTP 1.0 ad libitum for 5 days in confinement
  Arms: CHTP 1.0
Other: Conventional Cigarette (CC) — Subject's own preferred brand of CC ad libitum for 5 days in confinement
  Arms: Conventional cigarette (CC)

SUMMARY:
The overall goal of the study is to demonstrate the reduction of biomarkers of exposure (BoExp) to selected harmful and potentially harmful constituents (HPHCs) in adult smokers switching for 5 days from conventional cigarette (CC) to Carbon Heated Tobacco Product 1.0 (CHTP 1.0) as compared to smokers continuing to use CC.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥ 21 years.
* Subject is Caucasian.
* Subject is healthy, as judged by the Investigator.
* Subject smokes at least 10 commercially available non-menthol CCs per day (no brand restrictions) for at least the last 6 weeks prior to admission, based on self-reporting.
* Subject has smoked at least for the last 3 years.
* Subject does not plan to quit smoking in the next 3 months.

Exclusion Criteria:

* As per Investigator judgment, the subject cannot participate in the study for any reason (e.g., medical, psychiatric, and/or social reason).
* Subject has received medication within 14 days or within 5 half-lives of the medication (whichever is longer), which has an impact on cytochrome P450 1A2 (CYP1A2) or cytochrome P450 2A6 (CYP2A6) activity.
* Female subject is pregnant or breast feeding.
* Female subject does not agree to use an acceptable method of effective contraception.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christelle Haziza, PhD, Study Chair — Philip Morris Products S.A.; Katarzyna Jarus-Dziedzic, MD, PhD, Principal Investigator — BioVirtus Research Site
Locations (1):
- BioVirtus Research Site Sp. z o.o., Kajetany, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tran CT, Bosilkovska M, de La Bourdonnaye G, Blanc N, Haziza C. Reduced levels of biomarkers of exposure in smokers switching to the Carbon-Heated Tobacco Product 1.0: a controlled, randomized, open-label 5-day exposure trial. Sci Rep. 2020 Nov 5;10(1):19227. doi: 10.1038/s41598-020-76222-y. PMID 33154508

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study initiated (first subject screened): 04 July 2015
  At admission (Day -3), all the subjects performed a product trial of the CHTP 1.0. During the baseline period, they continued smoking their single preferred brand of CC. Then, on Day -1, subjects were randomized to one of the two study arms (CHTP 1.0 or CC) in a 1:1 ratio.
Pre-assignment Details: Enrolled and randomized population = 80 subjects
  * 41 subjects in CHTP 1.0 arm
  * 39 subjects in CC arm
  Number of subjects enrolled but NOT randomized (who tried the CHTP 1.0 at Day -3) = 5
Period: Overall Study
Arm/Group | CHTP 1.0 | Conventional Cigarette (CC)
Started | 41 | 39
Completed | 41 | 39
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study population consisted of all the randomized subjects who had at least 1 post randomization product use experience (CHTP 1.0 or CC), and at least 1 valid non-safety assessment.
  80 randomized subjects: 41 in CHTP 1.0 and 39 in CC study arms. All the randomized subjects completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | CHTP 1.0 | Conventional Cigarette (CC) | Total
Number analyzed (Participants) | 41 | 39 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (10.45) | 32.7 (10.97) | 33.5 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 20 | 19 | 39
International Organization for Standardization (ISO) nicotine level [Count of Participants; unit: Participants]
  ≤ 0.6 mg | 32 | 34 | 66
  > 0.6 to ≤ 1 mg | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Monohydroxybutenyl Mercapturic Acid (MHBMA)
Description: Concentrations measured on Day 5 in urine, adjusted for creatinine.
  Geometric Least Squares (LS) means are provided as descriptive statistics.
Time Frame: 5 days
Population: The analysis was performed on the full analysis set (FAS) population.
  The FAS consisted of all the randomized subjects who had at least 1 post randomization product use experience (CHTP 1.0 or CC) and had at least 1 non-safety assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | CHTP 1.0 | Conventional Cigarette (CC)
Number analyzed (Participants) | 41 | 39
pg/mg creat | 327.08 [282.39 to 378.84] | 1903.61 [1637.48 to 2212.99]
Statistical Analysis 1: Comparison: CHTP 1.0 vs Conventional Cigarette (CC); The hypothesis to be tested is that the geometric mean level on Day 5 of the biomarker of exposure for CHTP 1.0 is lower relative to CC. Analysis of the BoExp was conducted on the natural log scale in order to test the following hypothesis (one sided test with 2.5% type I error probability): * Null hypothesis (H0): m1≥m2 * Alternative hypothesis (H1): m1<m2 Where m1 and m2 are the geometric means of the BoExp levels on Day 5 for CHTP 1.0 and CC, respectively; Test type: Superiority or Other; p < .001, ANCOVA — The primary endpoints were tested using a multiple testing procedure to preserve the overall alpha level by simultaneously testing the endpoints using a closed procedure with each test performed at a two-sided alpha level of 5%; ANCOVA model on MHBMA levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Reduction = 82.82, 95% CI 2-sided [78.79 to 86.09] — Geometric LS Mean Reduction = 100 - (CHTP 1.0 : CC ratio) Expressed as %

2. Primary Outcome: Concentration of 3-hydroxypropylmercapturic Acid (3-HPMA)
Description: Concentrations measured on Day 5 in urine, adjusted for creatinine.
  Geometric Least Squares means are provided as descriptive statistics.
Time Frame: 5 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mg creat
Arm/Group | CHTP 1.0 | Conventional Cigarette (CC)
Number analyzed (Participants) | 41 | 39
ng/mg creat | 464.27 [432.13 to 498.80] | 1272.96 [1182.66 to 1370.15]
Statistical Analysis 1: Comparison: CHTP 1.0 vs Conventional Cigarette (CC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model on 3-HPMA levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Reduction = 63.53, 95% CI 2-sided [59.55 to 67.12] — Geometric LS Mean Reduction = 100 - (CHTP 1.0 : CC ratio) Expressed as %

3. Primary Outcome: Concentration of S-phenylmercapturic Acid (S-PMA)
Description: as for outcome 2
Time Frame: 5 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mg creat
Arm/Group | CHTP 1.0 | Conventional Cigarette (CC)
Number analyzed (Participants) | 41 | 39
pg/mg creat | 352.39 [321.26 to 386.54] | 2971.98 [2703.14 to 3267.55]
Statistical Analysis 1: Comparison: CHTP 1.0 vs Conventional Cigarette (CC); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < .001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA model on MHBMA levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Reduction = 88.14, 95% CI 2-sided [86.46 to 89.62] — Geometric LS Mean Reduction = 100 - (CHTP 1.0 : CC ratio) Expressed as %

4. Primary Outcome: Levels of Carboxyhemoglobin (COHb)
Description: % COHb blood measurements performed in the evening of Day 5, expressed as % of saturation of hemoglobin.
  Geometric Least Squares means are provided as descriptive statistics.
Time Frame: 5 days
Population: The analysis was performed on the full analysis set (FAS) population: all randomized subjects who had at least 1 post randomization product use experience (CHTP 1.0 or CC) and had at least 1 non-safety assessment.
  However, due to sample issues such as clotting, COHb assessment results could not be generated for some of the subjects.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of saturation of hemoglobin
Arm/Group | CHTP 1.0 | Conventional Cigarette (CC)
Number analyzed (Participants) | 32 | 26
percentage of saturation of hemoglobin | 2.660 [2.316 to 3.054] | 6.460 [5.531 to 7.544]
Statistical Analysis 1: Comparison: CHTP 1.0 vs Conventional Cigarette (CC); The hypothesis to be tested is that the geometric mean level on Day 5 of the biomarker of exposure for CHTP 1.0 is lower relative to CC. Analysis of the BoExp was conducted on the natural log scale in order to test the following hypothesis (one sided test with 2.5% type I error probability): * Null hypothesis (H0): m1≥m2 * Alternative hypothesis (H1): m1<m2 Where m1 and m2 are the geometric means of the BoExp levels on Day 5 for CHTP 1.0 and CC respectively; Test type: Superiority or Other; p < .001, ANCOVA — The primary endpoints were tested using a multiple testing procedure to preserve the overall alpha level by simultaneously testing the endpoints using a closed procedure with each test performed at an alpha level of 2.5% one sided; ANCOVA model on COHb levels with product, sex, cigarette consumption, and baseline value as covariates; Geometric LS Mean Ratio = 58.83, 95% CI 2-sided [49.30 to 66.56] — Geometric LS Mean Reduction = 100 - (CHTP 1.0 : CC ratio) Expressed as %

ADVERSE EVENTS:
Time Frame: From the informed consent form signature until the end of the safety follow-up period, up to 58 days (including a screening period of up to 42 days, a 9-day confinement period followed by a 7-day safety follow-up period (7 days after discharge of the subject or early discontinuation)).
Description: The safety was assessed in the safety population, consisting of 85 subjects: 80 randomized subjects (41 in CHTP 1.0 and 39 in CC) and 5 subjects exposed to CHTP 1.0 during the product trial on Day -3 but not randomized.
Groups:
- Enrolled But Not Randomized: Subjects who tried the CHTP 1.0 at Admission (Day -3) but were not randomized
Arm/Group | CHTP 1.0 | Conventional Cigarette (CC) | Enrolled But Not Randomized
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/39 | 1/5
Other Adverse Events (participants affected / at risk) | 27/41 | 14/39 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHTP 1.0 (N=41) | Conventional Cigarette (CC) (N=39) | Enrolled But Not Randomized (N=5)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Concussion was considered to be moderate in intensity and not related to the CHTP 1.0 or CC but to study procedures. This serious adverse event was considered to have resolved after 4 days. The subject had no ongoing medical conditions at Screening
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHTP 1.0 (N=41) | Conventional Cigarette (CC) (N=39) | Enrolled But Not Randomized (N=5)
Headache (Nervous system disorders) | 19 (21) | 9 (13) | 3 (3)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (17) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vessel puncture site haematoma (General disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specifies that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belongs to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2015-06-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT02503254/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT02503254/SAP_001.pdf